CLINICAL TRIAL: NCT04574622
Title: Effect of Session Frequency of Radial Extracorporeal Shock Wave Therapy (rESWT) on Gastrocnemius Muscle Spasticity in Children With Spastic Type Cerebral Palsy: A Double-Blinded, Randomized Clinical Trial
Brief Title: Effect of Session Frequency of rESWT on Gastrocnemius Muscle Spasticity in Children With Spastic Type Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rizky Kusuma Wardhani (Other)
Responsible Party: Sponsor-Investigator, Rizky Kusuma Wardhani, M.D., Physiatrist, Consultant in PM&R Department, Indonesia University
Organization: Indonesia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KET885/UN2F1/ETIK/PPM0002/2019
Record Dates: First submitted 2020-09-22; First posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Spasticity, Muscle; Cerebral Palsy; Child; Spastic
Keywords: Spasticity; Cerebral Palsy; Children; ESWT; Frequency
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants (including parents of patients), physiatrists who conducted ESWT and physiatrists who examined the patients' ASAS score are all blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Five true ESWT sessions (Experimental): A total of five sessions (1x/week) were conducted.
  A total of 1,500 pulses were delivered to each gastrocnemius muscle. The energy flux density was constant at 0.1 mJ/mm2 and the repetition frequency was at 4 Hz, with a pressure of 1.5 bars.
  Interventions: Device: radial Extracorporeal Shockwave Therapy
- Three true ESWT sessions and two sham ESWT sessions (Experimental): A total of three true ESWT (week 1, 3 and 5) and two sham ESWTs in (week 2 and 4) were conducted.
  For true ESWT sessions, a total of 1,500 pulses were delivered to each gastrocnemius muscle. The energy flux density was constant at 0.1 mJ/mm2 and the repetition frequency was at 4 Hz, with a pressure of 1.5 bars.
  For sham ESWT sessions, a total of 1,500 pulses were delivered to each gastrocnemius muscle with a 1 cm gap between between the probe and subject's skin. The energy flux density was constant at 0.1 mJ/mm2 and the repetition frequency was at 4 Hz, with a pressure of 1.5 bars.
  Interventions: Device: radial Extracorporeal Shockwave Therapy

INTERVENTIONS:
Device: radial Extracorporeal Shockwave Therapy — rESWT was given on gastrocnemius muscles with the subject lying on prone position. No anesthesia was required.

SUMMARY:
Spasticity, defined as a velocity dependent increase in tonic stretch reflexes, is one of the most prominent motor problems that occur in patients with cerebral palsy (CP). This causes difficulty in achieving balance, mobility, and an upright stance. CP is a group of permanent disorders that affect the development of movement and posture caused by a non-progressive damage to the brain. Because CP occurs in 2-3 of 1000 individuals, it is one of the most common causes of severe physical disability in children.

Mismanagement of spasticity can lead to contracture which is extremely difficult to treat and may result in severe functional disabilities. The current management of spasticity in CP includes physical therapy (i.e. passive stretching), oral medication, botulinum toxin injection, and surgery. Botulinum toxin injection has been proven to effectively reduce spasticity yet many patients are unable to get access to this treatment due to its high cost. Moreover, Botulinum toxin injection is currently not covered by the public health insurance of Indonesia. Therefore, other modalities which are more affordable and are non-invasive therapies should be considered as a treatment option for spasticity.

Radial Extracorporeal Shockwave Therapy (rESWT) has been utilized in the medical practice for the treatment of several musculoskeletal disorders such as chronic tendinopathies and spasticity. It is hypothesized that ESWT has two main effects which include a direct effect from mechanical forces at the treatment point and an indirect effect from cavitation. Even though rESWT has less penetration capacity over the focused Extracorporeal Shockwave Therapy (fESWT), rESWT is still believed to be more superior to fESWT because it requires less precise focusing, is less painful, and costs less. These also make rESWT the more appropriate choice for children with CP.

Many studies have proven the efficacy of ESWT in reducing spasticity in spastic CP patients with significantly long lasting effects. Despite promising results, there still has yet to be a recommended guideline for the treatment of spasticity in children using rESWT. One of the critical parameters needed to be determined is the frequency of treatment. Therefore, the objective of this study is to understand whether the reduction in gastrocnemius stiffness in children with spastic CP is influenced by the frequency of ESWT sessions.

DETAILED DESCRIPTION:
This study was designed as a double-blinded and randomized controlled trial.

Pediatric CP patients from the Department of Physical Medicine and Rehabilitation at Rumah Sakit Umum Pusat Nasional Dr. Cipto Mangunkusumo (RSCM) are involved in this research. Participants were selected using the inclusion criteria as follow: 1) children with spastic CP who are 5 - 18 years old, 2) one or two gastrocnemius muscle with an Australian Spasticity Assessment Scale (ASAS) of two or more, 3) at least 6 months since the last botulinum injection on gastrocnemius, 4) no surgical operation on lower limb within the last 12 months, 5) absence of severe contracture on gastrocnemius, and 6) ability of legal caregiver to provide written informed consent.

The spasticity of gastrocnemius was evaluated using ASAS (0: no spasticity to 4: severe spasticity). Data were collected at nine time points: 1) pre-ESWT, 2-6) immediately after each ESWT session, 7) 4 weeks after the last (fifth) ESWT session, 8) 8 weeks after the last (fifth) ESWT session, and 9) 12 weeks after the last (fifth) ESWT session. All patients were examined by the same physiatrist who was blinded to the protocol (i.e. not informed about the study and the group allocation) throughout the whole study.

The investigators used a BTL-6000 SWT Topline (BTL, Czech Republic) to apply rESWT on gastrocnemius muscles. For the procedures, a 1.2 cm probe was used. A total of 1,500 pulses were delivered to each gastrocnemius muscle. The energy flux density was constant at 0.1 mJ/mm2 and the repetition frequency was at 4 Hz, with a pressure of 1.5 bars.

For double-blinded treatment, 28 different spastic gastrocnemius muscles from 14 CP patients were allocated into two groups. Both groups had a true or sham ESWT for five consecutive weekly treatments. Group I received five true ESWT sessions. Group II received three true ESWT in session 1, 3 and 5 and two sham ESWTs in session 2 and 4. No anesthesia was given. Adverse events were closely monitored during and after therapy.

Intra-group changes in ASAS were evaluated with Friedman analysis of variance from baseline, immediately after each ESWT, 4 weeks after last (fifth) ESWT, 8 weeks after last (fifth) ESWT and 12 weeks after last (fifth) ESWT; followed by post-hoc Wilcoxon signed-ranked test. Inter-group differences in ASAS reduction were analyzed using Mann-Whitney U- test. Statistical analysis was conducted using SPSS ver. 23.0 (IBM Corporation, Armonk, NY, USA). The level of significance was set at <0.05.

ELIGIBILITY:
Inclusion Criteria:

* patients with spastic CP aged 5 to 18 years old
* at least one gastrocnemius with an Australian Spasticity Assessment Scale (ASAS) of 2 or more
* ability of legal respondent to give written informed consent

Exclusion Criteria:

* 6 months or less since the last botulinum injection on hamstring
* surgical operation on lower limb within the last 12 months
* severe contracture on gastrocnemius

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-06-17 (Actual); Study Completion 2020-06-17 (Actual)

PRIMARY OUTCOMES:
Baseline Spasticity of Gastrocnemius | pre-ESWT
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)
Spasticity of Gastrocnemius after first ESWT session | After first ESWT session (Week 1)
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)
Spasticity of Gastrocnemius after second ESWT session | After second ESWT session (Week 2)
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)
Spasticity of Gastrocnemius after third ESWT session | After third ESWT session (Week 3)
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)
Spasticity of Gastrocnemius after fourth ESWT session | After fourth ESWT session (Week 4)
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)
Spasticity of Gastrocnemius after fifth ESWT session | After fifth ESWT session (Week 5)
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)
Spasticity of Gastrocnemius four weeks after fifth (last) ESWT session | Four weeks after fifth (last) ESWT session (Week 9)
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)
Spasticity of Gastrocnemius eight weeks after fifth (last) ESWT session | Eight weeks after fifth (last) ESWT session (Week 13)
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)
Spasticity of Gastrocnemius twelve weeks after fifth (last) ESWT session | Twelve weeks after fifth (last) ESWT session (Week 17)
  Evaluated as the degree of resistance to passive movement using ASAS (0: no spasticity to 4: severe spasticity)

CONTACTS AND LOCATIONS:
Overall Officials: Rizky K Wardhani, M.D., Physiatrist, Principal Investigator — Universitas Indonesia Fakultas Kedokteran
Locations (1):
- Universitas Indonesia Fakultas Kedokteran, Jakarta Pusat, DKI Jakarta, Indonesia